CLINICAL TRIAL: NCT04777968
Title: Evaluation Of Fluoride Uptake By Dentine Following Pretreatment With Silver Diamine Fluoride And Potassium Iodide Under Resin Modified Glass Ionomer Restoration Versus Resin Modified Glass Ionomer Restoration Alone In Carious Primary Molars: (In Vitro Study)
Brief Title: Evaluation Of Fluoride Uptake By Dentine Following Silver Diamine Fluoride Under Resin Modified Glass Ionomer Restoration In Carious Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Associate Professor Dr. Rania Abdallah Nasr, Associate Professor Dr. Rania Nasr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19739
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
Keywords: Silver Diamine Fluoride; Resin Modified Glass Ionomer; Fluoride Uptake; Carious primary teeth
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: Extracted Discarded Primary Molars divided into CONTROL Group & INTERVENTIONAL Group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principle investigator & co-investigator are masked before assessing the outcomes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (A) : RMGI restoration without SDF and KI. (No Intervention): • RMGI restoration without SDF and KI.
- Intervention Group (B): Pretreatment with SDF and KI prior to RMGI restoration. (Experimental): • Pretreatment with SDF and KI prior to RMGI restoration.
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — a layer of 38% SDF solution was topically applied to the cavity using a micro brush, immediately followed by a saturated Potassium Iodide KI solution using a micro brush also, then a creamy white precipitate was immediately formed, KI was applied until the white precipitate turned clear.
  Other Names: SDF and KI
  Arms: Intervention Group (B): Pretreatment with SDF and KI prior to RMGI restoration.

SUMMARY:
Dental caries is one of the most common oral diseases of childhood and is considered as a major public health problem especially in areas with poor access to dental care. In a recent cross sectional study carried out in Egypt on 1000 child aged from 3-6 years, it was found that 61.4% of these children had dental caries. In order to avoid serious complications of untreated dental caries such as pain, infections, emergency visits and possibly hospitalization , an effective low cost treatment should be identified particularly in areas with poor dental access.

Studies have proven that silver diamine fluoride (SDF) is a topical fluoride that has the ability to effectively arrest and prevent dental caries.

DETAILED DESCRIPTION:
It was concluded that fluoride uptake into dentine from conventional GI restorations was not affected in the presence of SDF and KI. It was also mentioned that the results may be different if conditioning is applied not etching and recommended this for future investigation.

Aim: Therefore, the aim of this study is to determine whether carious primary molars treated with SDF and Potassium iodide (KI) prior to placing resin modified glass ionomer (RMGI) restorations will affect the fluoride uptake into primary dentine or not.

Study Setting:

* The study was conducted in Pediatric Dentistry and Dental Public Health Department Faculty of Dentistry, Cairo University, Egypt.
* Energy Dispersive X-ray analysis with Scanning Electron Microscope (SEM/EDX) measurement analysis was conducted at the National Research Center (NRC), Egypt.

Freshly extracted discarded primary molars were collected from outpatient clinic of Pediatric Dentistry Department, Faculty of Dentistry, Cairo University at the end of every day.

* Teeth were then sectioned through the center of the carious lesion mesiodistally using a slow-speed cutting saw with coolant (Isomet 4000, USA) forming two similar halves, so that the 20 molars were sectioned to 40 halves.
* Each tooth was placed in a separate container with its 2 halves.
* Teeth containers were then randomly allocated either to the control or intervention group.

Control Group: One half empty and the other half with Resin Modified Glass Ionmer (RMGI) only.

Intervention Group : One half empty and the other half SDF+KI+RMGI

* After dehydration, teeth were mounted on stubs using double-sided carbon tape, and sputter coated with gold for 20 s using a Turbo molecular pumped coater (QUORUM 150T ES, Laughton, United Kingdom) .
* Teeth were then placed in SEM/EDX for fluoride measurement by weight percentage.

Data showed parametric distribution so; it was represented by mean and standard deviation (SD) values. Independent and paired t-tests were used for inter and intragroup comparisons respectively. The significance level was set at p ≤0.05 within all tests. Statistical analysis was performed with R statistical analysis software version 4.0.3 for windows (R Core Team, 2020).

ELIGIBILITY:
Inclusion Criteria:

* • Carious primary extracted molars.

  * Presence of occlusal or proximal caries.
  * Caries extending to dentine.

Exclusion Criteria:

* • Presence of restorations.

  * Presence of pit and fissure sealant.
  * Hypolpastic teeth.
  * Severly destructed teeth. Thirty two teeth were collected, but only 20 teeth were eligible according to the inclusion and exclusion criteria. Teeth were then stored in distilled water

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Fluoride uptake into dentine | 2 weeks
  Fluoride weight percent in dentin under Resin Modified Glass Ionomer Restoration in primary molars

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Assoc. Prof., Principal Investigator — Faculty of Dentistry, Cairo University, Egypt
Locations (2):
- Egypt (2):
  - Department of Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo
  - Faculty of Dentistry, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No
Protocol and Abstract